CLINICAL TRIAL: NCT03180944
Title: Lower Lugol's Solution Concentration on Reducing the Adverse Symptoms of Chromoendoscopy With Iodine Staining
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2017SDU-QILU-G001
Record Dates: First submitted 2017-06-04; First posted 2017-06-08 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Mucosal Irritation; Image Quality
Keywords: Lugol's solution; esophageal squamous cell cancer; mucosal irritation; image quality
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Lugol's solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1.2% Lugol's solution (Experimental): This group patients were given concentrations of 1.2% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 1.2% Lugol's solution
- 1.0% Lugol's solution (Experimental): This group patients were given concentrations of 1.0% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 1.0% Lugol's solution
- 0.8% Lugol's solution (Experimental): This group patients were given concentrations of 0.8% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 0.8% Lugol's solution
- 0.6% Lugol's solution (Experimental): This group patients were given concentrations of 0.6% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 0.6% Lugol's solution
- 0.4% Lugol's solution (Experimental): This group patients were given concentrations of 0.4% Lugol's solution for chromoendoscopy.
  Interventions: Drug: 0.4% Lugol's solution

INTERVENTIONS:
Drug: 1.2% Lugol's solution — This group patients were given concentrations of 1.2% Lugol's solution for chromoendoscopy.Then biopsy specimens will be taken at the well-demarcated unstained or less-stained lesions.
  Arms: 1.2% Lugol's solution
Drug: 1.0% Lugol's solution — This group patients were given concentrations of 1.0% Lugol's solution for chromoendoscopy.Then biopsy specimens will be taken at the well-demarcated unstained or less-stained lesions.
  Arms: 1.0% Lugol's solution
Drug: 0.8% Lugol's solution — This group patients were given concentrations of 0.8% Lugol's solution for chromoendoscopy.Then biopsy specimens will be taken at the well-demarcated unstained or less-stained lesions.
  Arms: 0.8% Lugol's solution
Drug: 0.6% Lugol's solution — This group patients were given concentrations of 0.6% Lugol's solution for chromoendoscopy.Then biopsy specimens will be taken at the well-demarcated unstained or less-stained lesions.
  Arms: 0.6% Lugol's solution
Drug: 0.4% Lugol's solution — This group patients were given concentrations of 0.4% Lugol's solution for chromoendoscopy.Then biopsy specimens will be taken at the well-demarcated unstained or less-stained lesions.
  Arms: 0.4% Lugol's solution

SUMMARY:
This study was to test an optimal concentration of Lugol's solution which can reduce the mucosal irritation and provide high image quality to ensure endoscopy examination by a randomized blinded controlled trial.

DETAILED DESCRIPTION:
It is widely accepted that chromoendoscopy using Lugol's solution is effective for the detection of early esophageal squamous neoplasia. However, this modality may cause severe chest pain and discomfort owing to mucosal irritation. The conventional concentration of Lugol's solution is in the range of 1.2% to 2.5% . Image quality can be guaranteed with this range of Lugol's solution. However, lead to retrosternal pain and discomfort, and can even induce erosion or ulceration in the esophagus and stomach. This study was to test whether a lower concentration of Lugol's solution, which has minimal mucosal irritation, can provide satisfied image quality by a randomized blinded controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients in the high-risk population of ESCC;
* or general risk population of ESCC between 40 to 74 years old. Definition of high-risk population of ESCC is list in supporting information33.

Exclusion criteria included the following:

* with obvious abnormalities in stomach, confirmed by either white-light endoscopy (WLE) or pCLE, including gastric cancer, acute erosive and hemorrhagic gastritis, chronic atrophic gastritis, H. pylori infection and severe bile reflux gastritis;
* advanced esophageal carcinoma;
* known esophageal surgery or endoscopic treatment;
* known esophageal radiotherapy or chemotherapy;
* esophageal stenosis;
* food retention;
* allergy to iodine or fluorescein sodium;
* hyperthyroid;
* coagulopathy;
* acute bleeding;
* severe organ failure;
* pregnant or breastfeeding women.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Image Quality | intraoperative
  Image quality is blindly quantified by a 4-point scale from the endoscopists. A higher score representing higher image quality.

SECONDARY OUTCOMES:
Gastric Mucosa Injury | 1 months
  The gastric mucosal injury caused by Lugol's solution is defined as post-staining gastritis score minus pre-staining gastritis score in pCLE. The confocal gastritis was graded 0 to 3,according to pit patterns, capillaries, and fluorescein leakage. A higher score representing more serious injury.
Adverse Events | 24 hours
  Both a written and oral form of the Numerical Rating Scale (NRS) was provided to the patients after the endoscopy examination, used for measuring patients' retrosternal pain, retrosternal discomfort, nausea, abdominal discomfort and others. In NRS, 0 is painless, 10 is the most severe pain, less than 4 is mild pain (pain does not affect sleep), 4-6 is moderate pain, and more than 7 is severe pain (pain means unable to sleep or wake up from sleep).
Severe Adverse Events | 24 hours
  Severe adverse events includes allergic reactions, esophageal burns, spasms and even perforation.
Tolerance | intraoperative
  The 4-point scale was used to assess the tolerance of endoscopist to the esophageal spasm caused by Lugol's solution which prevent endoscopy from passing. 1-4 means the resistance as intolerable, tolerable, mild, or non-existing.
Histology analysis | 3-5days
  All specimens were evaluated by two experienced pathologists blind to the groups of the patients. The macroscopic and histologic diagnosis were made based on Paris classification and Vienna classification, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Qu JY, Li Y, Liu GQ, Li Z, Zhong N, Zhang MM, Li YY, Yu T, Lu XF, Li LX, Liu H, Qi QQ, Li YQ, Zuo XL. Optimal concentration of Lugol's solution for detecting early esophageal carcinoma: A randomized controlled trial. J Gastroenterol Hepatol. 2023 Jun;38(6):962-969. doi: 10.1111/jgh.16190. Epub 2023 Apr 24. PMID 37094943